CLINICAL TRIAL: NCT04206410
Title: Evaluation of the Effectiveness of Probiotics Stabilized With Cryoprotection Technology in Patients With Irritable Bowel Syndrome - a Randomized Double-blind, Placebo-controlled Study
Brief Title: Effectiveness of Probiotics Stabilized With Cryoprotection Technology in Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Memorial Health Institute, Poland (Other)
Collaborators: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Bożena Cukrowska, Principal Investigator, Children's Memorial Health Institute, Poland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6/KBE/2018
Record Dates: First submitted 2019-12-12; First posted 2019-12-20 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome, probiotics
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Probiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Multistrain probiotic mixture consisting of two Lactobacillus strains (L. rhamnosus and L. acidophilus) and three Bifidobacterium strains (B. longum, B. bifidum and B. lactis) administered for 8 weeks in a dose 1,0E+10/day, 2x sachets/day (5,0E+9/cfu per sachet)
  Interventions: Dietary Supplement: Probiotic
- Maltodextrin (Placebo Comparator): Placebo - Maltodextrin manufactured with an appearance, taste and packaging (sachets) identical to the probiotic mixture administarted for 8 weeks 2x sachets/day
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Probiotic — Multispecies probiotic mixture administered to patients according to the randomization list
  Arms: Probiotic
Dietary Supplement: Maltodextrin — Maltodextrin as placebo
  Arms: Maltodextrin

SUMMARY:
Irritable bowel syndrome (IBS) is one of the most common diseases of the digestive tract in adults, which pathogenesis is not fully understood. It is assumed that intestinal dysbiosis affecting the functioning of the gut-brain axis may be important. Probiotics are live microorganisms that, when administered at the right dose, have a positive effect on human health. Probiotic mechanism of action is related to the modulation of intestinal microbiota. Clinical studies confirm that probiotics administered to patients with IBS have positive health effects. Clinical effects depend primarily on the selection of probiotic strains, but no less important is their viability and stability in the preparation administered to patients. Unfortunately, obtaining stability (a strictly defined number of live probiotic strains in the preparation throughout the shelf life of the preparation) is very technologically difficult. As shown by the audit of the Polish Supreme Audit Office (NIK), almost 90% of probiotics sold on the Polish market do not meet these criteria. There were probiotic preparations that by the end of their expiration date had less than 100 live bacterial cells from the declared number of about one billion. The only preparations that successfully passed NIK inspections turned out to be preparations in which the technology of double microcapsulation of bacteria was used. New technologies are constantly being sought that increase both the survival of bacterial strains in the preparation and the resistance of the strains to hydrochloric acid and bile, which in turn contributes to delivering the right dose of probiotics to the target site of activity, i.e. the small and large intestine. Recent developed an innovative technology called bacterial cryoprotection, which, compared to traditional lyophilization, leads to an increase in the stability of the bacterial cell wall membranes and protects them against negative factors both external (high temperature, humidity etc.) and internal (gastric acid, bile). Therefore, the purpose of the clinical trial is to assess the effectiveness of cryoprotected probiotics in patients with IBS.

DETAILED DESCRIPTION:
A 1- to 2-week screening period will be used to establish the presence and persistence of trial entry criteria and train patients in the mode of data collection. The screening period will also be used to select patients with specified levels of severity of signs and symptoms. During screening visit patients will undergo physical examination. Severity of IBS will be determined using the Francis, Morris and Whorwell's IBS severity scale (IBS-SSS): Mild <175, Moderate 175-300, Severe >300. Number and type of stools will be measured in all patients using Bristol stool scale. All eligible patients who sign informed consent form will be randomized within 2 weeks to receive either probiotic product or placebo and will complete Quality of Life assessment measured using IBS-QOL questionnaire. They will also be instructed to restrain from consuming foods and dietary supplements containing probiotics according to the clinical study requirements. After receiving probiotic product/placebo, telephone interviewers will call patients 3 times per week, and they will collect the following information by the phone: type of stools (according to Bristol Stool Score), number of bowel movements per day and IBS symptoms measured in 5-point scale (abdominal pain, flatulence, feeling of incomplete evacuation). In addition, telephone interviewers will collect information regarding adverse effects and using new drugs during the study. Patients will report to the doctor 2 times during study every 4 weeks during 8 week lasting intervention to receive new dose of probiotic product/placebo and to be assessed by the doctor using IBS-SSS, IBS-GIS and IBS-AR questionnaires, They will also complete Quality of Life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects of Caucasian race
2. Age between 16 and 60 years (inclusive)
3. Good physical, medical and mental status estimated on the basis of the medical history and a general clinical examination.
4. Results of laboratory tests (hematology, clinical chemistry, serology, and urinalysis) within the normal range of the local laboratory or considered non-clinically significant by the investigator.
5. Subjects who have provided freely their own written informed consent.
6. Subjects available for the whole study period.
7. Diagnosed with diarrhea-predominant irritable bowel syndrome (IBS-D) according to Rome III criteria, i.e. symptoms of recurrent abdominal pain or discomfort* and a marked change in bowel habit with symptoms experienced on at least three days a week of at least three months within last year. Pain/discomfort is related to a change in the appearance of stool, frequency of stool and improves with defecation.

   * "Discomfort" means an uncomfortable sensation not described as pain.
8. The following subjects will be enrolled in the study:

   1. with diarrhea-predominant irritable bowel syndrome, i.e., persons, who have at least one stool of type 6 or type 7 in Bristol stool score (BSS) over at least 2 days a week
   2. with at least moderate form assessed using IBS-SSS (5 questions, maximum number of points 500); enrolled subjects with score >175 points Mild <175 points, Moderate 175-300 points, Severe >300 points.
9. Subjects who are able to follow strictly the instructions of the investigational team regarding the study procedures and to fulfil the requirements of the protocol.
10. The following medications are permitted during the course of the study, as long as they are used at a constant dosage and are commenced at least 1 month prior to study start:

    1. birth control pill, or depot intramuscular contraceptive preparation,
    2. estrogen-progesterone replacement therapy,
    3. L-thyroxine,
    4. low-dose antidepressants (up to 25 mg day of amitriptyline, nortriptyline, or selective serotonin reuptake inhibitor)
    5. low-dose antihypertensives in the diuretic, angiotensin-converting enzyme inhibitor or angiotensin II inhibitor classes.

Exclusion Criteria:

1. Patients with cardiovascular disorders: uncontrolled hypertension (blood pressure > 170/100 mmHg), cerebrovascular diseases.
2. Patients with respiratory disorders (asthma, chronic obstructive pulmonary disease [COPD]).
3. Patients with hepatic disorders (including condition following cholecystectomy procedure) and renal disorders as well as abnormal results of biochemical blood tests without diagnosis: serum creatinine > 2 x upper limit of normal, AST or ALT > 2 x upper limit of normal.
4. Patients with gastrointestinal disorders other than IBS, including clinically or endoscopic-confirmed gastroenteritis.
5. Patients with endocrinological disorders, including patients with diabetes mellitus (fasting blood glucose concentration > 11 mmol/L), and TSH > normal.
6. Patients with serious neurological disorders, psychosis.
7. Patients with malignancies.
8. Pregnant or lactating women.
9. Soy hypersensitivity.
10. The subject has been diagnosed with lactose intolerance and this can explain their symptoms (i.e., symptoms resolved or reduced significantly with lactose-free diet).
11. Use of motility drugs or dietary fiber supplements within 2 weeks before study start.
12. Patients, taking anti-coagulant medication.
13. Plan to have surgery during the time of the study.
14. Currently consuming probiotics and refuse to have a three months washout period.
15. Recent antibiotic therapy within the last 3 month.
16. Patients, who receive antibiotics during the study, will be excluded.
17. Patients, enrolled in another clinical trial in the past 3 months.
18. The subject has a history of alcohol or substance abuse.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Improvement or worsening of IBS global symptoms using Global Improvement Scale (IBS-GIS) | Improvement/worsening of global symptoms after 4 and 8 weeks of intervention
  IBS-Global Improvement Scale asseses IBS symptoms using a patient-defined 7 point Linkert scale ranging from symptoms substantially worse to substantially improved.
  Patients answer the question "Have you felt any change in the severity of your symptoms over the past 7 days compared to how you felt before the medicine was given?
  The answers are recorded based on the 7-point scale:
  1. = I feel that the symptoms have worsened significantly
  2. = I feel that the symptoms have moderately worsened
  3. = I feel that the symptoms have slightly worsened
  4. = I feel no change
  5. = I feel a slight improvement
  6. = I feel moderate improvement
  7. = I feel significant improvement
  IBS-GIS score indicates: improvement if is >4 or worsening if is<4, no change if is 4
Changes in severity of IBS symptoms using IBS Severity Scoring System (IBS-SSS) | From baseline at 4 and 8 weeks of intervention
  IBS-Severity Scoring System is a 5-question survey that asks: 1. the severity of abdominal pain, 2. frequency of abdominal pain, 3. severity of abdominal distention, 4.dissatisfaction with bowel habit, and 5. interference with quality of life over the past 10 days. Subjects respond to each question on a 100-point visual analogue scale. Each of the five question generates a maximum score of 100 point, and total scores can range from 0-500 with higher scores indicating severe symptoms. A decrease of 50 points is associated with a clinically meaningful improvement.
Changes in adequate relief of IBS symptoms (IBS-AR) | From baseline at 4 and 8 weeks of interventions
  IBS-Adequate Relief (IBS-AR) is a dichotomous single item that asks participants "Over the past week (7 days) have you had adequate relief of your IBS symptoms? The answer is YES or NO.
Changes in Quality of Life (IBS-QOL) | From baseline at 4 and 8 weeks of intervention
  The IBS-Quality of Life (IBS-QOL) is a 34-item measure assessing the degree to which IBS interferes with patient quality of life. Each item is rated on a 5-point Likert scale, thus yielding a total score that has a theoretical range of 34 to 170, with higher scores indicating worse QOL.

SECONDARY OUTCOMES:
Changes in type of stools | From baseline for 8 weeks of intervention
  Type of stool assessed before intervention and then 3 times a week. Type of stools assessed using the Bristol Stool Scale. Bristol Scale is designed to classify faeces into seven groups: type 1-2 indicate constipation, type 3-4 are "normal" stools; type 5-7 indicate diarrhea.
Changes in severity of pain | From baseline for 8 weeks of intervention
  The severity of pain assessed before intervention and then 3 times a week using a patient-defined 5 point Linkert scale: point 0 - no pain, and 1-4 the severity of pain with higher scores indicating worse pain.
Changes in flatulence | From baseline for 8 weeks of intervention
  The severity of flatulence assessed before intervention and then 3 times a week using a patient-defined 5 point Linkert scale: point 0 - no flatulence, and points1-4 with higher scores indicating worse flatulence
Changes in feeling of incomplete evacuation of stool | From baseline for 8 weeks of intervention
  The severity of incomplete evacuation of stool assessed before intervention and then 3 times a week using a patient-defined 5 point Linkert scale: point 0 - no feeling of incomplete evacuation of stool, and points1-4 with higher scores indicating worse feeling of incomplete evacuation of stool
Changes in number of bowel movements per day | From baseline for 8 weeks of intervention
  Number of bowel movements per day assessed before intervention and then 3 times a week.

OTHER OUTCOMES:
Changes in serum level of intestinal fatty acid binding protein | From baseline at 8 weeks of intervention
  Intestinal fatty acid binding protein (I-FABP) is a novel serological marker of disrupted enterocytes, and could be an indicator of increased intestinal permeability. The level is measured in patients' sera using commercially available kits.

CONTACTS AND LOCATIONS:
Overall Officials: Bożena Cukrowska, PhD MD, Principal Investigator — The Children's Memorial Health Institute
Locations (1):
- The Children's Memorial Health Institute, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skrzydlo-Radomanska B, Prozorow-Krol B, Cichoz-Lach H, Majsiak E, Bierla JB, Kosikowski W, Szczerbinski M, Gantzel J, Cukrowska B. The Effectiveness of Synbiotic Preparation Containing Lactobacillus and Bifidobacterium Probiotic Strains and Short Chain Fructooligosaccharides in Patients with Diarrhea Predominant Irritable Bowel Syndrome-A Randomized Double-Blind, Placebo-Controlled Study. Nutrients. 2020 Jul 5;12(7):1999. doi: 10.3390/nu12071999. PMID 32635661